CLINICAL TRIAL: NCT06373224
Title: Evaluating the Use of Preventive Cold Saline to Decrease Bleeding Associated With Endobronchial Biopsy
Brief Title: Cold Saline Irrigation Before Endobronchial Biopsy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23-037
Record Dates: First submitted 2023-08-03; First posted 2024-04-18 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Lung Diseases
Keywords: Biopsy
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flush Group (Experimental): After identifying the lymph node or lesion to be biopsied on ultrasound, using the endobronchial ultrasound scope, two 60mL syringes of cold saline will be inserted, through the biopsy channel of the endobronchial ultrasound scope, directly onto the bronchial wall where the biopsies are to be performed. The saline will then be sucked out of the airway using the endobronchial ultrasound scope.
  Interventions: Other: Flush
- Standard Care Group (No Intervention): No irrigation before the biopsy

INTERVENTIONS:
Other: Flush — After identifying the lymph node or lesion to be biopsied on ultrasound, using the endobronchial ultrasound scope, two 60mL syringes of cold saline will be inserted, through the biopsy channel of the endobronchial ultrasound scope, directly onto the bronchial wall where the biopsies are to be performed. The saline will then be sucked out of the airway using the endobronchial ultrasound scope.
  Arms: Flush Group

SUMMARY:
Patients undergoing an endobronchial ultrasound and biopsy can experience bleeding during the biopsy. These biopsies are read in real time by pathologists who travel to the endoscopy unit during the procedure. Often, when this happens, the blood contaminates the pathology slides making the slide unreadable. This then requires more biopsies to be performed, thus prolonging the procedure, and increasing anesthesia time. One innovative way to reduce bleeding may be to irrigate the bronchial wall with cold saline, where the biopsy is to be taken, immediately before biopsy, thus causing vasoconstriction and possibly resulting in less blood contamination on the biopsy slides. The current study will evaluate this prophylactic irrigation with saline to control bleeding, thus resulting in a quicker diagnostic result of the biopsies.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing an endobronchial ultrasound and biopsy at Bethesda North Hospital

Exclusion Criteria:

* Under 18 years old
* Does not speak English
* Unable to consent to involvement in the research study
* Is pregnant
* Has a bleeding disorder/diagnosis
* Currently taking anticoagulant medications and not stopped for procedure
* Documented low platelets (<100,000)
* Had a biopsy taken immediately prior to the endobronchial ultrasound

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-12-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of unreadable biopsy slides | from enrollment until discharge from biopsy appointment, up to 12 hours
  Number of biopsy slides noted by the pathologist to be unreadable due to blood on slide

CONTACTS AND LOCATIONS:
Overall Officials: Austin Pittman, BSN, RN, Principal Investigator — TriHealth Inc.
Locations (1):
- Bethesda North Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No